CLINICAL TRIAL: NCT00035477
Title: Efficacy and Safety of Azimilide for the Treatment of Patients With Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Preston M Dunnmon, MD, Procter & Gamble Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000038
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — azimilide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo tablets in hospital and placebo tablets outpatient
  Interventions: Drug: Placebo
- 2 (Experimental): Azimilide tablets in hospital and azimilide tablets outpatient
  Interventions: Drug: Azimilide Dihydrochloride

INTERVENTIONS:
Drug: Azimilide Dihydrochloride — 125 mg azimilide tablets once a day for 3 days in hospital and 125 mg azimilide tablets once a day for 6 months as outpatient
  Arms: 2
Drug: Placebo — placebo tablets once a day for 3 days in hospital and placebo tablets once a day for 6 months as outpatient
  Arms: 1

SUMMARY:
Atrial fibrillation (abnormal rhythm in the upper chamber of the heart) is a common supraventricular arrhythmia (abnormal heart rhythm) for which antiarrhythmic therapy is often prescribed. The primary goals of therapy are to maintain sinus rhythm (normal heart rhythm) and to reduce the occurrence of episodes of atrial fibrillation. Azimilide may have an effect on increasing the time to first recurrence of symptomatic atrial fibrillation or atrial flutter and symptomatic paroxysmal supraventricular tachycardia (other types of abnormal heart rhythms).

This double-blind, placebo-controlled study is designed to evaluate the efficacy and safety of azimilide compared with placebo in maintaining sinus rhythm in patients who require cardioversion (electric shock to correct heart rhythm) to reduce atrial fibrillation. Once this phase of the study is completed, a second phase with a different study design will be conducted. The second phase is an open-label follow-up phase to the study. This follow-up phase will continue to evaluate the long-term efficacy and safety of a daily oral dose of azimilide in patients who complete the double-blind, placebo-controlled phase of this study.

ELIGIBILITY:
Inclusion criteria:

* Documented (12-lead ECG) history of symptomatic atrial fibrillation occurring between 48 hours and 6 months before screening
* Require the procedure of cardioversion (electric shock to correct heart rhythm)
* In the investigator's opinion, be likely to maintain sinus rhythm after cardioversion.
* Be anticoagulated according to the recommendations of the Study Group on Atrial Fibrillation of the European Society of Cardiology guidelines.

Exclusion criteria:

* Previously unsuccessful electrical cardioversions
* Failed to respond to any Class III antiarrhythmic drugs
* Qualifying arrhythmia due to acute reversible illness, acute myocardial infarction, and/or cardiac or thoracic surgery within one month prior to randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2000-09; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Prolong the time from start of teh efficacy period to the first symptomatic or asymptomatic event fo AFIB, etc | six months

CONTACTS AND LOCATIONS:
Overall Officials: Preston M Dunnmon, MD, Study Director — Procter and Gamble
Locations (82):
- United States (69):
  - The Heart Group, PC, Mobile, Alabama
  - University Medical Center, Tucson, Arizona
  - Cardiovascular Associates of Penisula, Burlingame, California
  - San Diego Cardiovascular Research Associates, Encinitas, California
  - La Mesa Cardiac Center, a Medical Group, La Mesa, California
  - Good Samaritan Hospital, Los Angeles, California
  - LAC + USC Medical Center, Los Angeles, California
  - Cardiology Section, West Los Angeles VA Hospital, Los Angeles, California
  - Merced Heart Associates, Merced, California
  - Sutter Gould Medical Foundation, Modesto, California
  - ARI Clinical Trials, Redondo Beach, California
  - Inland Clinical Research, Riverside, California
  - Regional Cardiology Assoc., Sacramento, California
  - Cardiology Associates, San Diego, California
  - Western Cardiology Assoc., Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The George Washington University MFA, Washington D.C., District of Columbia
  - Cardiology Consultants, Daytona Beach, Florida
  - C/O Research Office Attn: Cardiovascular Research Dept., Fort Lauderdale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Lakeland Regional Medical, Lakeland, Florida
  - Khalid Hasan Sheikh 80 Fortenberry Road, Merritt Island, Florida
  - Florida Cardiology, Orlando, Florida
  - Cardiology Reasearch Assiocates, Ormond Beach, Florida
  - VA Medical Center, Decatur, Georgia
  - Elgin Cardiology Associates, Elgin, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Heart Center Medical Group, Fort Wayne, Indiana
  - The Care Group, Indianapolis, Indiana
  - University of Louisville-Cardiology, Louisville, Kentucky
  - Louisville Cardiology Medical Group, P.S.C., Louisville, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Richard Gilmore 501 S. Ryan Street, Lake Charles, Louisiana
  - Cardiovascular Instiute of the South, Morgan City, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Androscoggin Cardiology Associates Research, Auburn, Maine
  - Maine Medical Center, Portland, Maine
  - University of Massachusett, Worcester, Massachusetts
  - Thoracic & Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Riverside Osteopathic Hospital, Trenton, Michigan
  - Regional Heart Center, Duluth, Minnesota
  - VA Medical Center Therapeutic Section, Minneapolis, Minnesota
  - St. Paul Heart Clinic, Saint Paul, Minnesota
  - Duke Medical Center, Durham, North Carolina
  - Altru Health System Research Center, Grand Forks, North Dakota
  - Lindner Clinical Trial Ctr., Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Hillsboro Cardiology, Hillsboro, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Heart Care Group PC, Allentown, Pennsylvania
  - Tri-State Medical Group Cardiology, Beaver, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Pavillion, Jenkintown, Pennsylvania
  - UPHS/Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Cardiovascular and Critical Care Associates, P.C., Pittsburgh, Pennsylvania
  - Cardiology Foundation of Lankenau, Wynnewood, Pennsylvania
  - Charleston Cardiology, Charleston, South Carolina
  - Stern Cardiovascular Center Research Department, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Heart and Vascular Inst. of Texas, PA, San Antonio, Texas
  - Riverside Regional Medical Center, Newport News, Virginia
  - Daniel Gottlieb 16259 Sylvester Road SW Suite 401, Seattle, Washington
  - FHS Research, Tacoma, Washington
  - Beloit Clinic, SC, Beloit, Wisconsin
  - Wisconsin Center for Clinical Research, Elkhorn, Wisconsin
  - Dean/Riverview Clinic, Janesville, Wisconsin
  - University of Wisconsin Madison, Madison, Wisconsin
  - Wisconsin Center for Clinical Research, Milwaukee, Wisconsin
- Canada (13):
  - University of Calgary, Calgary, Alberta
  - Rockyview General Hospital CV Lab Research, Calgary, Alberta
  - Cardiology Research St. Paul's Hospital, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Neureka Research Corporation, Greater Sudbury, Ontario
  - Hamilton Health Sciences Crop, Hamilton, Ontario
  - Cardiac Investigation Unit, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Recherche Cardiologie, Montreal, Quebec
  - Hospital Sacre-Coeur de Montreal, Montreal, Quebec
  - Quebec Heart Institute, Sainte-Foy, Quebec